CLINICAL TRIAL: NCT00483678
Title: A Pilot Study of an Intimacy-Enhancing Couples Therapy for Men With Advanced Prostate Cancer and Their Partners
Brief Title: Couples Therapy to Enhance Intimacy Between Patients With Advanced or Recurrent Prostate Cancer and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 07-043; P30CA008748 (NIH); MSKCC-07043
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Sexual Dysfunction; Sexuality and Reproductive Issues
Keywords: psychosocial effects of cancer and its treatment; sexual dysfunction; sexuality and reproductive issues; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Sexuality | interventions — Counseling; Psychiatric Rehabilitation

ARMS (2):
- Intimacy-Enhancing Couples Therapy (Experimental): Patients and their partners receive Intimacy-Enhancing Couples Therapy over 6 weeks comprising the following four 90-minute sessions: the Story of Cancer; Understanding the Couple, Ways of Relating and Key Influences; Intimacy; and Coping, Support, and Adaptation. Patients and their partners complete treatment satisfaction questionnaires after completion of study intervention.
  Interventions: Other: counseling intervention; Other: questionnaire administration; Procedure: psychosocial assessment and care
- standard psychosocial care (Active Comparator): Patients and their partners receive standard psychosocial care. All participants complete questionnaires assessing psychological distress, intimacy, communication patterns, and overall relationship adjustment/satisfaction at baseline and at 1 month after completion of study intervention
  Interventions: Other: questionnaire administration; Procedure: psychosocial assessment and care

INTERVENTIONS:
Other: counseling intervention
  Arms: Intimacy-Enhancing Couples Therapy
Other: questionnaire administration
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: A couples therapy program may enhance intimacy and reduce psychological distress in patients with prostate cancer and in their partners.

PURPOSE: This randomized clinical trial is studying how well couples therapy enhances intimacy and reduces psychological distress in patients with advanced or recurrent prostate cancer and in their partners.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of Intimacy-Enhancing Couples Therapy (IECT) for patients with advanced or recurrent prostate cancer and their partners.
* Compare the effect of IECT vs usual care on patients' and their partners' level of global psychological distress.
* Compare the effect of IECT vs usual care on relationship intimacy in these participants.

OUTLINE: This is a randomized, controlled, pilot, multicenter study. Patients are stratified according to marital distress based on partners' scores on the Abbreviated Dyadic Adjustment Scale (high [< 21] vs low [≥ 21]). Patients and their partners are randomized to 1 of 2 arms.

* Arm I: Patients and their partners receive Intimacy-Enhancing Couples Therapy over 6 weeks comprising the following four 90-minute sessions: the Story of Cancer; Understanding the Couple, Ways of Relating and Key Influences; Intimacy; and Coping, Support, and Adaptation. Patients and their partners complete treatment satisfaction questionnaires after completion of study intervention.
* Arm II: Patients and their partners receive standard psychosocial care. All participants complete questionnaires assessing psychological distress, intimacy, communication patterns, and overall relationship adjustment/satisfaction at baseline and at 1 month after completion of study intervention.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary prostate cancer

  * Advanced or recurrent disease
* Receiving concurrent hormonal therapy
* Married and/or co-habitating with a partner for ≥ 1 year
* T-score > 50 on Brief Symptom Inventory-18 questionnaire (patient and/or partner)

PATIENT CHARACTERISTICS:

* Normal cognitive functioning
* Able to speak and read English
* No significant hearing impairment that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intimacy-Enhancing Couples Therapy (IECT) (e.g., eligibility rate, acceptance rate, attendance rate, satisfaction) assessed at baseline and at 1 month after completion of study intervention | 2 years
Comparison of the preliminary effect of IECT vs usual care on global psychological distress and relationship intimacy as assessed by the BSI-18 at baseline and at 1 month after completion of study intervention | 2 years
Relationship functioning, including intimacy, communication, and satisfaction (cancer-specific and overall) as assessed by the CRCS and A-DAS at baseline and at 1 month after completion of study intervention | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Talia Zaider, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center - Cheltenham, Philadelphia, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/